CLINICAL TRIAL: NCT03293771
Title: Assessment of Postoperative Urologic and Pelvic Floor Complaints in Male-to-female Transgender Patients: a Mixed Methods Study
Brief Title: Transgender Post-reassignment Urogynecologic Measures and Perceptions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); The Cleveland Clinic (Other); Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1708018495
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Gender Identity Disorder of Adult; Voiding Disorders; Sexual Dysfunction
Keywords: Transgender women; Male-to-female; Gender confirmation surgery; Voiding disorder; Vaginal dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage 1 Focus Groups: The focus groups will involve transgender women who have completed gender confirmation surgery who volunteer to discuss their postoperative experience regarding bladder function, genital complaints, and sexual function.
  Interventions: Other: Focus group interviews
- Stage 2 Questionnaire Groups: Stage 2 participants will be asked to complete a questionnaire packet after surgery followed by a second questionnaire completion 2 weeks later. Participants' operative notes and postoperative visit records will be reviewed.
  Interventions: Diagnostic Test: Questionnaire packet

INTERVENTIONS:
Other: Focus group interviews — Focus group participants will be asked about their postoperative urogynecologic experience. Confidentiality will be enforced and participants will be made aware that they may opt out of answering any questions.
  Groups: Stage 1 Focus Groups
Diagnostic Test: Questionnaire packet — Participants will be asked to complete a questionnaire packet comprised of three previously validated questionnaires and one newly created focused questionnaire. They will be asked to complete the new questionnaire again 2 weeks later. We estimate about 10 minutes will be required to complete the packet.
  Groups: Stage 2 Questionnaire Groups

SUMMARY:
The intent of this mixed methods study for transgender women after gender confirmation surgery is to characterize and subsequently create a validated screening questionnaire for postoperative urologic and pelvic floor symptoms. For individuals who seek gender-confirming treatment, about 13% undergo genital surgery for cosmetic purposes with or without gonadectomy, and this number is increasing. Patient satisfaction following surgery is high, particularly regarding sexual and cosmetic outcomes; however, unexpected negative functional outcomes such as bowel and bladder dysfunction and pelvic organ prolapse impact overall patient satisfaction. The available information suggests that 16-33% of patients experience incontinence postoperatively, with stress predominance, 32-47% experience abnormal voiding, and 24-66% experience overactive bladder symptoms. Outside of the typically assessed voiding symptoms, unique complaints of MTF postoperative patients include obstructive voiding symptoms due to urethral stenosis, persistent perimeatal erectile tissue, prostatic hypertrophy, and irritation from neovaginal tissue. Additionally, may of these patients develop symptomatic neovaginal prolapse, requiring re-suspension. We suggest that further clarification regarding MTF postoperative urologic and pelvic floor complaints can be achieved via a mixed methods approach. By using focus group interviews to create specific evaluative questions for this unique population, we can then prospectively assess patients undergoing surgery via a national multicenter sampling strategy. The goal of the study is to better understand the unique symptoms these women experience and create a validated, reliable screening questionnaire to monitor patients after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1 -- Male-to-female transgender women who are at least 4 weeks postoperative following genital surgery for gender confirmation
* Stage 2 -- Male-to-female transgender women who are scheduled to undergo surgery or are within 4 weeks postoperative
* Both stages -- Minimum age 18 years old
* Both stages -- English fluency
* Both stages -- Reliable contact information and/or permanent residence

Exclusion Criteria:

* Preexisting pelvic pathology, including abnormal anatomy or baseline voiding dysfunction
* Urinary or intestinal problems prior to surgery lasting greater than 6 weeks

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study participants involve transgender individuals who were born phenotypically male but identify as female.
Study Population: Stage 1 (Focus group) participants will be comprised of healthy volunteers from the transgender community who have completed male-to-female gender confirmation surgery. They will be recruited through local clinics, physician referral, or community support groups.
  Stage 2 (Questionnaire) participants will be recruited through multiple transgender centers at time of surgical scheduling or within 4 weeks after male-to-female gender confirmation surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-12-27 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Focus groups | 3 months
  Characterization of genital, urologic, bowel, and sexual symptoms following male-to-female gender confirmation surgery
Stage 2: Questionnaire testing | 12 months
  Validity and reliability testing of new questionnaire

SECONDARY OUTCOMES:
Frequency and severity of symptoms | 15 months
  Frequency and severity of symptoms
Relationship between surgical technique and symptoms | 15 months
  Relationship between surgical technique and symptoms
Effect of hormonal therapy usage and symptoms | 15 months
  Effect of hormonal therapy usage and symptoms
Length of time since surgery and development of symptoms | 15 months
  Length of time since surgery and development of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Huber, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Selvaggi G, Bellringer J. Gender reassignment surgery: an overview. Nat Rev Urol. 2011 May;8(5):274-82. doi: 10.1038/nrurol.2011.46. Epub 2011 Apr 12. PMID 21487386
- [Background] Clements-Nolle K, Marx R, Katz M. Attempted suicide among transgender persons: The influence of gender-based discrimination and victimization. J Homosex. 2006;51(3):53-69. doi: 10.1300/J082v51n03_04. PMID 17135115
- [Background] Kailas M, Lu HMS, Rothman EF, Safer JD. PREVALENCE AND TYPES OF GENDER-AFFIRMING SURGERY AMONG A SAMPLE OF TRANSGENDER ENDOCRINOLOGY PATIENTS PRIOR TO STATE EXPANSION OF INSURANCE COVERAGE. Endocr Pract. 2017 Jul;23(7):780-786. doi: 10.4158/EP161727.OR. Epub 2017 Apr 27. PMID 28448757
- [Background] Revol M, Servant JM, Banzet P. [Surgical treatment of male-to-female transsexuals: a ten-year experience assessment]. Ann Chir Plast Esthet. 2006 Dec;51(6):499-511. doi: 10.1016/j.anplas.2006.02.006. Epub 2006 Apr 19. French. PMID 16626849
- [Background] Hess J, Rossi Neto R, Panic L, Rubben H, Senf W. Satisfaction with male-to-female gender reassignment surgery. Dtsch Arztebl Int. 2014 Nov 21;111(47):795-801. doi: 10.3238/arztebl.2014.0795. PMID 25487762
- [Background] Goddard JC, Vickery RM, Qureshi A, Summerton DJ, Khoosal D, Terry TR. Feminizing genitoplasty in adult transsexuals: early and long-term surgical results. BJU Int. 2007 Sep;100(3):607-13. doi: 10.1111/j.1464-410X.2007.07017.x. PMID 17669144
- [Background] Buncamper ME, van der Sluis WB, van der Pas RSD, Ozer M, Smit JM, Witte BI, Bouman MB, Mullender MG. Surgical Outcome after Penile Inversion Vaginoplasty: A Retrospective Study of 475 Transgender Women. Plast Reconstr Surg. 2016 Nov;138(5):999-1007. doi: 10.1097/PRS.0000000000002684. PMID 27782992
- [Background] Jarolim L, Sedy J, Schmidt M, Nanka O, Foltan R, Kawaciuk I. Gender reassignment surgery in male-to-female transsexualism: A retrospective 3-month follow-up study with anatomical remarks. J Sex Med. 2009 Jun;6(6):1635-1644. doi: 10.1111/j.1743-6109.2009.01245.x. Epub 2009 Mar 30. PMID 19473463
- [Background] Rossi Neto R, Hintz F, Krege S, Rubben H, Vom Dorp F. Gender reassignment surgery--a 13 year review of surgical outcomes. Int Braz J Urol. 2012 Jan-Feb;38(1):97-107. doi: 10.1590/s1677-55382012000100014. PMID 22397771
- [Background] Hoebeke P, Selvaggi G, Ceulemans P, De Cuypere G, T'Sjoen G, Weyers S, Decaestecker K, Monstrey S. Impact of sex reassignment surgery on lower urinary tract function. Eur Urol. 2005 Mar;47(3):398-402. doi: 10.1016/j.eururo.2004.10.008. Epub 2004 Dec 2. PMID 15716207
- [Background] Lawrence AA. Patient-reported complications and functional outcomes of male-to-female sex reassignment surgery. Arch Sex Behav. 2006 Dec;35(6):717-27. doi: 10.1007/s10508-006-9104-9. Epub 2006 Nov 16. PMID 17109225
- [Background] Horbach SE, Bouman MB, Smit JM, Ozer M, Buncamper ME, Mullender MG. Outcome of Vaginoplasty in Male-to-Female Transgenders: A Systematic Review of Surgical Techniques. J Sex Med. 2015 Jun;12(6):1499-512. doi: 10.1111/jsm.12868. Epub 2015 Mar 26. PMID 25817066
- [Background] Kuhn A, Santi A, Birkhauser M. Vaginal prolapse, pelvic floor function, and related symptoms 16 years after sex reassignment surgery in transsexuals. Fertil Steril. 2011 Jun;95(7):2379-82. doi: 10.1016/j.fertnstert.2011.03.029. Epub 2011 Apr 2. PMID 21458798
- [Background] Kuhn A, Hiltebrand R, Birkhauser M. Do transsexuals have micturition disorders? Eur J Obstet Gynecol Reprod Biol. 2007 Apr;131(2):226-30. doi: 10.1016/j.ejogrb.2006.03.019. Epub 2006 May 5. PMID 16678333
- [Background] Dietrich W, Haitel A, Huber JC, Reiter WJ. Expression of estrogen receptors in human corpus cavernosum and male urethra. J Histochem Cytochem. 2004 Mar;52(3):355-60. doi: 10.1177/002215540405200306. PMID 14966202
- [Derived] Huber S, Ferrando C, Safer JD, Pang JHY, Streed CG Jr, Priestley J, Culligan P. Development and Validation of Urological and Appearance Domains of the Post-Affirming Surgery Form and Function Individual Reporting Measure (AFFIRM) for Transwomen following Genital Surgery. J Urol. 2021 Dec;206(6):1445-1453. doi: 10.1097/JU.0000000000002141. Epub 2021 Jul 21. PMID 34288738